CLINICAL TRIAL: NCT06873919
Title: A Geriatric Mobile Team for Nursing Home Residents: an Exploratory, Prospective, Single-Center, Non-Randomized, Non-Interventional Feasibility Pilot Study
Brief Title: A Geriatric Mobile Team for Nursing Home Residents: a Feasibility Pilot Study
Acronym: GerMoT
Status: Not yet recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: CHU UCL Namur (Unknown)
Responsible Party: Sponsor
Other Study IDs: GerMoT; 40025834 (Other: Fond National de la Recherche)
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nursing Home Resident; Geriatric Assessment
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental group: Nursing home resident with a geriatric consultation at her place of residence
  Interventions: Other: Geriatric assessment

INTERVENTIONS:
Other: Geriatric assessment — The tertiary hospital's geriatrics department is implementing a one-year mobile team composed of a geriatrician and a nurse to conduct geriatric assessments (Anamnesis and heteroanamnesis - Clinical examination - Medication review - Proposed management plan provided to the general practionner, who independently decides which recommendations to implement) in three nursing homes. This non-randomized pilot project aims to establish a new standard of care for residents selected by their primary care physician. The project is accompanied by a clinical study designed to assess the feasibility, effectiveness, and acceptability of this intervention. Prospectively collected data will also help define key indicators for a future large-scale study focusing on cost-effectiveness.

SUMMARY:
Nursing home (NH) residents have complex healthcare needs. Barriers to collaboration hinder the delivery of high-quality care in nursing homes. To bridge the gap between hospital-based and NH-based care, various innovative approaches have been proposed, including geriatric mobile teams. In Belgium, geriatric expertise has long been confined to hospital settings. Until recently, no specific organization existed for outpatient geriatric assessment, particularly for NH residents. In April 2024, the National Institute for Health and Disability Insurance (INAMI) introduced a new reimbursement code for geriatric consultations in NHs, promoting the development of extramural geriatric activities. However, evidence on the effectiveness of mobile geriatric teams remains limited, particularly regarding hospitalization prevention.

The geriatrics department of CHU UCL Namur is implementing a one-year pilot project involving a mobile team composed of a geriatrician and a nurse to conduct geriatric assessments in the three nursing homes. This non-randomized pilot project aims to establish a new standard of care for residents selected by their general practitioner, leveraging the new reimbursement code. The project is accompanied by a clinical study assessing the feasibility, effectiveness, and acceptability of this intervention. Prospectively collected data will also help define key indicators for a future large-scale study focused on cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 70 years
* Presenting with one or more of the following conditions:

  * Difficulties in establishing an advance care planning
  * Medical complexity (multiple specialists, repeated hospitalizations)
  * Polypharmacy
  * Recurrent falls
  * Unmanageable behavioral disorders
  * Weight loss
  * Memory impairment

Exclusion Criteria:

* Patients with an unstable medical condition requiring urgent care
* Patients under 70 years old
* Patients whose condition requires examinations or treatments available only in a hospital setting

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will be defined based on the population identified within the geriatric consultation project in nursing homes. Eligible patients present with geriatric syndromes identified by their primary care physician. They are over 70 years old and reside in one of the three nursing homes participating in the project.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasability | Immediately after the initial consultation, with follow-up assessments at 3, 6, 9, and up to 12 months post-inclusion.

SECONDARY OUTCOMES:
Acceptability | Immediately after the initial consultation, with follow-up assessments at 3, 6, 9, and up to 12 months post-inclusion
Determine the outcomes for a future full evaluation study. | Immediately after the initial consultation, with follow-up assessments at 3, 6, 9, and up to 12 months post-inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU UCL Namur, Yvoir, Belgium

IPD SHARING:
Plan to Share IPD: No